CLINICAL TRIAL: NCT05982067
Title: The Utility of MIndfulness-based Physical Exercise Program (MIPE Program) for Community-dwelling Older People With Sarcopenia: a Pilot Randomised Controlled Trial
Brief Title: MIndfulness-based Physical Exercise Program (MIPE Program) on Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Patrick KOR Pui Kin, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mindful PE Sarcope
Record Dates: First submitted 2023-07-07; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the character of the intervention and control group in this study (the mindfulness-based PE vs health education), it is impossible to blind participants. The interventionist (the qualified mindfulness instructor and sport coach) is also unrealizable to be blinded. To reduce the allocation bias as much as possible, the following personnel will be blinded: the research assistants who are responsible for the participants recruitment, the research assistants who perform the randomization and the assessor who collect data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness-based physical exercie (Experimental): The participants will receive about 70-min MIPE program twice a week, which will be conducted in a hybrid way, a combination of face-to-face and at home by a qualified mindfulness therapist and a sport coach.
  Interventions: Other: mindfulness-based phsycial exercise intervention
- Health education (Placebo Comparator): Health education consisting of discussion provided by a registered nurse will be conducted as a control of socialization and interaction.
  Interventions: Other: health education

INTERVENTIONS:
Other: mindfulness-based phsycial exercise intervention — The intervention is 12 weeks, two times a week. The MIPE intervention will be conducted in a hybrid way, a combination of face-to-face and at home, by a qualified mindfulness therapist and a qualified sport coach. Specifically, the participants will attend the face-to-face sessions once every two weeks and in other weeks, they will perform the intervention at home using videos and templates. The face-to-face sessions will be conducted at the health care centre. The intervention of each session will include 1) introduce the theme of this session, 2) mini lectures about the theme; 3) mindfulness practice related to the theme; 4) tips of keeping mindfulness during PE; 5) warm up: lead with mindfulness words; 6) resistance exercise; 7) cool down: lead with mindfulness words; 8) discussion.
  Arms: mindfulness-based physical exercie
Other: health education — The number of sessions, duration, frequency, group size and delivery modality will be similar to the intervention group. The topics of the health education are the care of common diseases in the older adults, including hypertension, diabetes, osteoporosis, COPD, dementia, depression. Each session is about 70 min (same as intervention group), including 10-20 min lecture and 50-60 discussion and sharing.
  Arms: Health education

SUMMARY:
The goal of this pilot randomized controlled trial (RCT) is to assess the feasibility, acceptability, and the preliminary effects of the MIndfulness-based Physical Exercise (MIPE) intervention among community-dwelling older people with sarcopenia. The main questions are: 1) is the MIPE intervention feasible and acceptable in older adults with sarcopenia? 2) is the MIPE intervention effective to improve the adherence to physical exercise intervention, alleviate the symptoms of sarcopenia and enhance the psychological well-being of older adults with sarcopenia? To answer these questions, a MIPE intervention protocol was developed by Delphi approach and end-users' evaluation. This pilot RCT will be conducted to assess the feasibility, acceptability, and the preliminary effects of the MIPE intervention. In the parallel-group, pilot RCT, 60 community-dwelling older people aged 60 years or older diagnosed with sarcopenia will be randomized into either the intervention group receiving the MIPE intervention 2 sessions weekly over 12 weeks or the control group receiving health educations. Each session of the MIPE intervention will last about 70 minutes, including 20-min mindfulness-based intervention, 40-min physical exercise (10-min warm-up, 20-min RE, and 10-min cool down) and 10-20-min sharing and discussion. The feasibility, acceptability and preliminary effectiveness on sarcopenia symptoms and psychological well-being of the MIPE program will be assessed.

DETAILED DESCRIPTION:
Background Sarcopenia is a geriatric syndrome characterised by low muscle mass, muscle strength, and physical function. Physical exercise (PE), especially resistance exercise, has demonstrated potential effects on sarcopenia. However, low motivation for regular PE is always reported as a major barrier in this population. Based on the PRIME (Plans, Responses, Impulses, Motives, and Evaluations) theory of motivation, Plan (i.e., well-planned, and evidence-based PE protocol), Motives (anticipated pleasure, satisfaction, and relief) and self-awareness on the present moment are the key points of human motivation and the potential targets to change a behaviour (i.e., adhering to a PE intervention) in older people with sarcopenia. Limited study on sarcopenia consisted of any interventional element to emphasise motives and self-awareness on the present moment, two key points of human motivation in the PRIME theory of motivation, although older people with sarcopenia are more likely to have negative feelings (i.e., fatigue, depress, anxiety) and experiences (i.e., derailed by daily life and distracted by concerns on PE). Mindfulness-based intervention (MBI) is a psychosocial intervention which aims to increase the participants' awareness of the present moment non-judgmentally. Increased evidence has indicated that MBI can also improve the levels of PE and adherence to PE interventions. Based on the mindful coping model, the positive relationship between mindfulness and PE might be that MBI has the potential to improve motivation for PE by addressing three key points of human motivation in the PRIME theory of motivation (focusing on the present moment, evoking positive feelings, and increasing self-awareness). Thus, MBI has the potential to be integrated into PE training to increase motivation and adherence to PE in older people with sarcopenia.

To address the above research gaps, we first conducted a SR on the home-based interventions among community-dwelling older people with sarcopenia was conducted, showing that home-based resistance exercise is feasible, suitable and has potential effects on sarcopenia, but few studies consisted of motivation-enhancing component. Then a Delphi study was conducted to develop the MIndfulness-based Physical Exercise (MIPE) intervention on this population. However, the feasibility, acceptability, and effects of the HOME intervention among community-dwelling older people with sarcopenia need to be explored.

Objective The objective of this study is to assess the feasibility, acceptability, and the preliminary effects of the MIPE intervention among community-dwelling older people with sarcopenia.

Methods A pilot randomised controlled trial (RCT) will be conducted to assess the feasibility, acceptability, and the preliminary effects of the HOME intervention. In the parallel-group, pilot RCT, 60 community-dwelling older people aged 60 years or older diagnosed with sarcopenia will be randomised into either the intervention group receiving the HOME intervention 2 sessions weekly over 12 weeks or the control group receiving health educations. Each session of the HOME intervention will last about 70 minutes, including 20-min MBI, 40-min HBE (10-min warm-up, 20-min RE, and 10-min cool down) and 10-20-min sharing and discussion. The feasibility of this programme will be determined by time spent recruiting participants, eligibility rate and recruitment rate. The acceptability of the HOME program will be assessed by: 1) prospective acceptability: recruitment rate and reasons for not involving in this study; 2) concurrent acceptability: attendance rate, complete rate, attrition rate and reasons for discontinuing; and 3) retrospective acceptability: the participants' perspectives on the intervention after taking part. Based on our conceptual framework, primary outcomes (muscle mass, muscle strength and physical function) and secondary outcomes (motivation, depressive symptoms, psychological well-being, mindfulness level and quality of life) will be assessed at baseline (T0), immediately post-intervention week 12 (T1) and 12 weeks after completion of the intervention. The quantitative data will be analysed by generalised estimating equations. The qualitative data will be Brun and Clark's thematic approach.

Impact and significance The MIPE program, consisting MBI and PE, is novel in the research field related to sarcopenia, which addresses the limitations of previous studies. This study has the potential to improve the symptoms of sarcopenia, the motivation and adherence to PE as well as the psychological health of this population, which finally improves the holistic welling of this population and facilitates their "ageing in place". For researchers, this study provides a relatively new sub-area in this field by generating insights on the importance of the above factors and the potential effectiveness of the mindfulness-based PE. For health professionals, the study provides a potentially effective way to improve the motivation and adherence to PE to treat sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling people aged 60 years or older
2. Diagnosed with sarcopenia by the criteria of the Asian Working Group for Sarcopenia (AWGS):

   1. decreased muscle strength: handgrip strength of males < 28 kg; handgrip strength of females < 18 kg;
   2. or decreased physical performance: the time of 5-time chair stand test ≥12 s;
   3. or decreased muscle mass: SMI of males is < 7.0 kg/m2; SMI of females is < 5.7 kg/m2
3. Able to communicate and written and understand the instruction

Exclusion Criteria:

1. Been hospitalized for more than 5 days in the preceding 3 months
2. Unable to have body composition test, such as having heart pacemaker, vascular stent, steel plates and nails in the body
3. Contraindications to exercise, such as severe musculoskeletal disorders, severe cardiovascular diseases or spinal nerve injury
4. Having regular exercise: 150-minute moderate-intensity activity or 75-minute vigorous-intensity activity per week, with each session lasting at least 10 min in the past 3 months based on self-reported time and a self-perceived intensity via Borg Scale
5. Practicing mindfulness/yoga for >45 min a week in the 6 months prior to recruitment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Time spent recruiting participants | baseline (T0)
  The time spent recruiting participants is the period from the first day of recruiting participants to the last day of recruiting participants. This outcome will help us understand the feasibility of the MIPE program. Specifically, shorter time spent recruiting participants roughly reflects the higher feasibility of the MIPE program.
Eligibility rate | baseline (T0)
  The eligibility rate will be calculated by the number of eligible participants/the number of screened participants. The higher eligibility indicates the more potential participants.
Recruitment rate | baseline (T0)
  The recruitment rate will be calculated by the number of participants recruited/ the number of eligible participants. The higher recruitment rate indicates the higher willingness of the eligible participants to join the MIPE program.
Attendance rate | week 12 (T1)
  The attendance rate will be calculated by the attended sessions of the participants/ all sessions. The higher attendance rate roughly indicates the higher involvement of the participants in the MIPE program.
Complete rate | week 12 (T1)
  The complete rate will be calculated by the sessions that finished at least 80% / all attended sessions. The higher complete rate indicates the actual involvement of the participants in the MIPE program.
Attrition rate | week 12 (T1)
  The attrition rate will be calculated by the number of participants dropped out total number of participants. If the participants engage in less than 80% of online sessions will be considered as attrition. The higher attrition rate indicates the lower participation in the MIPE program.
The participants' perspectives on the intervention | week 12 (T1)
  The participants' perspectives on the intervention will be explored by individual interviews. There are mainly five questions in the individual interviews: 1) Generally, what do you think of this intervention? 2) What do you think of the content of this intervention? 3) What do you think of the frequency, duration and delivery mode of this intervention? 4) How about your motivation to exercise? 5) What recommendations do you have for this intervention? The results will help us to further revise and improve the MIPE to be more tailored to the older adults with sarcopenia. The individual interviews will be conducted by the PhD student who has received rigor trained in qualitative study methods and engaged in individual interviews before and a professor who has rich experience in conducting individual interviews and is familiar with sarcopenia and mindfulness.

SECONDARY OUTCOMES:
Skeletal muscle mass index | baseline (T0) and week 12 (T1, immediately post-intervention)
  Skeletal muscle mass index (SMI) will be assessed by Bioelectrical impedance analysis (Inbody 270, Korea). The procedure of testing is below: before the test, the participants will be required to remove every item that might influence the test, such as metal keys, bank cards, mobile phones, from their body, and then take off their shoes and socks. Then, they will be instructed to stand straight on the detector with two hands holding the handles of the detector for about one minute. During the testing, they will be not allowed to talk, move, or laugh. Higher Skeletal muscle mass index (SMI) means the higher muscle mass. Comparisons of changes of skeletal muscle mass index (SMI) will be considered as follows: baseline (T0)- week 12 (T1).
The Chinese version of the Behavioral Regulation in Exercise Questionnaire-2 (C-BREQ-2) | baseline (T0) and week 12 (T1, immediately post-intervention)
  The Chinese version of the Behavioral Regulation in Exercise Questionnaire-2 (C-BREQ-2) assesses the motivation of the participants to exercise. The C-BREQ-2 is a self-report measure with 18-items and each item is rated on a 5-point Likert scale from 0 to 4, with a higher score indicating higher motivation to exercise. Comparison of change of the C-BREQ-2 will be considered as follows: baseline (T0)- week 12 (T1).
The Chinese version of the short form Geriatric Depression Scale (GDS-15) | baseline (T0) and week 12 (T1, immediately post-intervention)
  The Chinese version of the short form Geriatric Depression Scale (GDS-15) assesses the depressive symptoms of the participants. The score of GDS ranges 0-15 with each "no" answers of item 1,5,7 and 11 scoring 1 while the rest items scoring 1 with "yes" answers. The classification of depressive symptoms based on the score is: score 0-4: normal; score 5-8: mild depression; score 9-11: moderate depression; score 12-15: severe depression. Comparison of change of the Chinese version of the GDS-15 will be considered as follows: baseline (T0)- week 12 (T1).
The Chinese version of Raff's Psychological Well-being Scale (RPWS-C) | baseline (T0) and week 12 (T1, immediately post-intervention)
  The Chinese version of Raff's Psychological Well-being Scale (RPWS-C) assesses the psychological well-being of the participants. The RPWS-C has 24 items, and each item is rated from 1 (strongly disagree) to 6 (strongly agree), with higher score indicating higher psychological well-being. Comparison of change of the RPWS-C will be considered as follows: baseline (T0)- week 12 (T1).
The Chinese Version of the Physical Activity Scale for the Elderly (PASE-C) | baseline (T0) and week 12 (T1, immediately post-intervention)
  The Chinese Version of the Physical Activity Scale for the Elderly (PASE-C) assesses the physical activity level of the participants. The PASE-C, consisting of 10-items, is a self-reported scale to measure the occupational, household, and leisure activities for the last seven days. Higher score of the PASE-C indicates higher physical activity. Comparison of change of the PASE-C will be considered as follows: baseline (T0)- week 12 (T1).
The Chinese version of Five Facet Mindfulness Questionnaire (FFMQ-15-C) | baseline (T0) and week 12 (T1, immediately post-intervention)
  The Chinese version of Five Facet Mindfulness Questionnaire (FFMQ-15-C) assesses the mindfulness level of the participants. The FFMQ-15-C has 15 items and each item is rated on a 5-point Likert scale, ranging from1 = "never or very rarely true" to 5 = "very often or always true", with higher total scores indicating a higher degree of mindfulness. Comparison of change of the FFMQ-15-C will be considered as follows: baseline (T0)- week 12 (T1).
The Chinese version of Sarcopenia and Quality of life (SarQoL®) | baseline (T0) and week 12 (T1, immediately post-intervention)
  The Chinese version of Sarcopenia and Quality of life (SarQoL®) assesses the quality of life of the participants. The SarQoL® has 22 items with higher score indicating higher quality of life. Comparison of change of the SarQoL® will be considered as follows: baseline (T0)- week 12 (T1).
Handgrip strength | baseline (T0) and week 12 (T1, immediately post-intervention)
  Handgrip strength will be measured by Jamar dynamometer (Jamar, 563213, USA) and the method refers to the recommendation of American Society of Hand Therapists. Comparisons of changes of handgrip strength will be considered as follows: baseline (T0)- week 12 (T1).
5-times Chair stand test | baseline (T0) and week 12 (T1, immediately post-intervention)
  5-times Chair stand test reflects the physical function and is an indicator in the sarcopenia diagnosis. The participants will be invited to stand and sit from a chair (about 43 cm) five times and the time will be recorded. Short time of the test, better physical function. Comparisons of changes of 5-times Chair stand test will be considered as follows: baseline (T0)- week 12 (T1).

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Suzhou, Jiangsu, China

REFERENCES:
- [Background] Cruz-Jentoft AJ, Sayer AA. Sarcopenia. Lancet. 2019 Jun 29;393(10191):2636-2646. doi: 10.1016/S0140-6736(19)31138-9. Epub 2019 Jun 3. PMID 31171417
- [Background] Mayhew AJ, Amog K, Phillips S, Parise G, McNicholas PD, de Souza RJ, Thabane L, Raina P. The prevalence of sarcopenia in community-dwelling older adults, an exploration of differences between studies and within definitions: a systematic review and meta-analyses. Age Ageing. 2019 Jan 1;48(1):48-56. doi: 10.1093/ageing/afy106. PMID 30052707
- [Background] Cao L, Morley JE. Sarcopenia Is Recognized as an Independent Condition by an International Classification of Disease, Tenth Revision, Clinical Modification (ICD-10-CM) Code. J Am Med Dir Assoc. 2016 Aug 1;17(8):675-7. doi: 10.1016/j.jamda.2016.06.001. No abstract available. PMID 27470918
- [Background] Beaudart C, Zaaria M, Pasleau F, Reginster JY, Bruyere O. Health Outcomes of Sarcopenia: A Systematic Review and Meta-Analysis. PLoS One. 2017 Jan 17;12(1):e0169548. doi: 10.1371/journal.pone.0169548. eCollection 2017. PMID 28095426
- [Background] Peng TC, Chen WL, Wu LW, Chang YW, Kao TW. Sarcopenia and cognitive impairment: A systematic review and meta-analysis. Clin Nutr. 2020 Sep;39(9):2695-2701. doi: 10.1016/j.clnu.2019.12.014. Epub 2019 Dec 17. PMID 31917049
- [Background] Chang KV, Hsu TH, Wu WT, Huang KC, Han DS. Is sarcopenia associated with depression? A systematic review and meta-analysis of observational studies. Age Ageing. 2017 Sep 1;46(5):738-746. doi: 10.1093/ageing/afx094. PMID 28633395
- [Background] Cho HW, Chung W, Moon S, Ryu OH, Kim MK, Kang JG. Effect of Sarcopenia and Body Shape on Cardiovascular Disease According to Obesity Phenotypes. Diabetes Metab J. 2021 Mar;45(2):209-218. doi: 10.4093/dmj.2019.0223. Epub 2020 Jul 10. PMID 32662256
- [Background] Yang M, Liu Y, Zuo Y, Tang H. Sarcopenia for predicting falls and hospitalization in community-dwelling older adults: EWGSOP versus EWGSOP2. Sci Rep. 2019 Nov 27;9(1):17636. doi: 10.1038/s41598-019-53522-6. PMID 31776354
- [Background] Nakamura K, Yoshida D, Honda T, Hata J, Shibata M, Hirakawa Y, Furuta Y, Kishimoto H, Ohara T, Kitazono T, Nakashima Y, Ninomiya T. Prevalence and Mortality of Sarcopenia in a Community-dwelling Older Japanese Population: The Hisayama Study. J Epidemiol. 2021 May 5;31(5):320-327. doi: 10.2188/jea.JE20190289. Epub 2020 Oct 17. PMID 32507775
- [Background] Su Y, Hirayama K, Han TF, Izutsu M, Yuki M. Sarcopenia Prevalence and Risk Factors among Japanese Community Dwelling Older Adults Living in a Snow-Covered City According to EWGSOP2. J Clin Med. 2019 Feb 28;8(3):291. doi: 10.3390/jcm8030291. PMID 30823497
- [Background] Bruyere O, Beaudart C, Ethgen O, Reginster JY, Locquet M. The health economics burden of sarcopenia: a systematic review. Maturitas. 2019 Jan;119:61-69. doi: 10.1016/j.maturitas.2018.11.003. Epub 2018 Nov 12. PMID 30502752
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Hurst C, Robinson SM, Witham MD, Dodds RM, Granic A, Buckland C, De Biase S, Finnegan S, Rochester L, Skelton DA, Sayer AA. Resistance exercise as a treatment for sarcopenia: prescription and delivery. Age Ageing. 2022 Feb 2;51(2):afac003. doi: 10.1093/ageing/afac003. PMID 35150587
- [Background] Wu PY, Huang KS, Chen KM, Chou CP, Tu YK. Exercise, Nutrition, and Combined Exercise and Nutrition in Older Adults with Sarcopenia: A Systematic Review and Network Meta-analysis. Maturitas. 2021 Mar;145:38-48. doi: 10.1016/j.maturitas.2020.12.009. Epub 2020 Dec 31. PMID 33541561
- [Background] Yoshimura Y, Wakabayashi H, Yamada M, Kim H, Harada A, Arai H. Interventions for Treating Sarcopenia: A Systematic Review and Meta-Analysis of Randomized Controlled Studies. J Am Med Dir Assoc. 2017 Jun 1;18(6):553.e1-553.e16. doi: 10.1016/j.jamda.2017.03.019. PMID 28549707
- [Background] Li ML, Kor PP, Sui YF, Liu JY. Health maintenance through home-based interventions for community-dwelling older people with sarcopenia during and after the COVID-19 pandemic: A systematic review and meta-analysis. Exp Gerontol. 2023 Apr;174:112128. doi: 10.1016/j.exger.2023.112128. Epub 2023 Feb 21. PMID 36804363
- [Background] Reangsing C, Rittiwong T, Schneider JK. Effects of mindfulness meditation interventions on depression in older adults: A meta-analysis. Aging Ment Health. 2021 Jul;25(7):1181-1190. doi: 10.1080/13607863.2020.1793901. Epub 2020 Jul 15. PMID 32666805
- [Background] Goldberg SB, Tucker RP, Greene PA, Davidson RJ, Wampold BE, Kearney DJ, Simpson TL. Mindfulness-based interventions for psychiatric disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2018 Feb;59:52-60. doi: 10.1016/j.cpr.2017.10.011. Epub 2017 Nov 8. PMID 29126747
- [Background] Wang S, Yin H, Jia Y, Zhao L, Wang L, Chen L. Effects of Mind-Body Exercise on Cognitive Function in Older Adults With Cognitive Impairment: A Systematic Review and Meta-analysis. J Nerv Ment Dis. 2018 Dec;206(12):913-924. doi: 10.1097/NMD.0000000000000912. PMID 30507734
- [Derived] Li ML, Kor PP, Zhang ZY, Liu JY. Feasibility and preliminary effects of a mindfulness-based physical exercise (MBPE) program for community-dwelling older people with sarcopenia: A protocol for a parallel, two-armed pilot randomised controlled trial. PLoS One. 2024 Apr 18;19(4):e0302235. doi: 10.1371/journal.pone.0302235. eCollection 2024. PMID 38635544